CLINICAL TRIAL: NCT00583674
Title: A Randomized, Double Blind, Multi-Center, Phase 2 Study to Estimate the Efficacy and Evaluate the Safety and Tolerability of Cisplatin & Capecitabine (CX) in Combination With AMG 386 or Placebo in Subjects With Metastatic Gastric, Gastroesophageal Junction, or Distal Esophageal Adenocarcinoma
Brief Title: Phase 2 Study of AMG 386 (20060439) in Combination With Cisplatin & Capecitabine in Subjects With Metastatic Gastric, Gastroesophageal Junction, or Distal Esophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060439
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastric Cancer; Metastatic Gastric, Gastroesophageal Junction, or Distal Esophageal Adenocarcinoma; AMG 386; Cisplatin; Capecitabine
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms | interventions — trebananib; Cisplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- B (Experimental)
  Interventions: Drug: AMG 386 3mg/kg; Drug: Cisplatin; Drug: Capecitabine
- A (Experimental)
  Interventions: Drug: AMG 386 10mg/kg; Drug: Cisplatin; Drug: Capecitabine
- C (Active Comparator)
  Interventions: Drug: AMG 386 placebo; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: AMG 386 placebo — AMG 386 placebo IV QW until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: C
Drug: AMG 386 10mg/kg — AMG 386 10 mg/kg IV QW until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: A
Drug: AMG 386 3mg/kg — AMG 386 3 mg/kg IV QW until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: B
Drug: Cisplatin — Cisplatin 80 mg/m2 IV Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: C
Drug: Capecitabine — Capecitabine1000 mg/m2 PO BID x 14 days Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: C
Drug: Cisplatin — Cisplatin 80 mg/m2 IV Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: A
Drug: Capecitabine — Capecitabine 1000 mg/m2 PO BID x 14 days Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: A
Drug: Cisplatin — Cisplatin 80 mg/m2 IV Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: B
Drug: Capecitabine — Capecitabine 1000 mg/m2 PO BID x 14 days Q3W until radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death
  Arms: B

SUMMARY:
This is a phase 2, randomized, double blind, placebo controlled, multi-center study to estimate the improvement in progression free survival (compared to control subjects) and evaluate the safety and tolerability of AMG 386 in combination with Cisplatin & Capecitabine in the treatment of subjects with Metastatic Gastric, Gastroesophageal Junction, or Distal Esophageal Adenocarcinoma. AMG 386 is a man-made medication that is designed to stop the development of blood vessels in cancer tissues. Cancer tissues rely on the development of new blood vessels, a process called angiogenesis, to obtain a supply of oxygen and nutrients to grow.

ELIGIBILITY:
Inclusion Criteria:

* Disease Related

  * Histologically or cytologically confirmed adenocarcinoma of the stomach, gastroesophageal junction or distal esophagus with metastatic disease
  * Measurable or non-measurable disease per RECIST Guidelines
  * Prior gastrectomy (total or partial) may be allowed as long as subjects can take oral medications and meet all other inclusion/exclusion criteria. Subjects may not take crushed or dissolved capecitabine via a feeding/gastrostomy tube
  * Palliative radiotherapy for metastatic esophageal or gastric cancer prior to study entry may be allowed as long as all toxicities from radiotherapy have resolved and the radiotherapy was not to the only site of known metastatic disease
* Demographic

  •18 years of age or older at the time the written informed consent is obtained
* General

  * Able to swallow oral medication
  * ECOG performance status of 0 or 1
* Laboratory

  * Adequate organ and hematological function as evidenced by laboratory studies prior to randomization

Exclusion Criteria:

* Disease Related

  * Prior chemotherapy for metastatic disease (1st line)
  * Less than 12 months have elapsed from completion of previous adjuvant or neoadjuvant chemotherapy or chemoradiotherapy
  * Subjects with persistent gastric outlet obstruction, complete dysphagia or feeding jejunostomy
  * Radiotherapy ≤ 14 days prior to randomization. Subjects must have recovered from all radiotherapy-related toxicities
  * Current or prior history of central nervous system metastases
  * History of arterial or deep venous thromboembolism within 12 months prior to randomization
  * History of bleeding diathesis or clinically significant bleeding within 6 months prior to randomization
  * Major surgical procedure within 28 days prior to randomization
  * Minor surgical procedure, placement of central venous access device or fine needle aspiration within 3 days prior to randomization
  * Prior malignancy except: malignancy treated with curative intent and without evidence of active disease for ≥ 3 years prior to randomization and felt to be at low risk for recurrence by treating physician, adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease, adequately treated cervical carcinoma in situ without evidence of disease, prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Prior malignancy (other than in situ cervical cancer, or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for ≥ 3 years prior to randomization
  * Clinically significant cardiovascular diseases within 12 months prior to randomization
  * Presence of clinically significant non-healing wound, ulcer (including gastrointestinal) or fracture as judged by the investigator
  * Ongoing or clinically significant active infection as judged by the investigator
  * Known hypersensitivity to bacterial proteins, or any of the drugs required in this study
  * Known peripheral neuropathy ≥Grade 1
  * Known dihydropyrimidine dehydrogenase deficiency
  * Known hypersensitivity to 5-FU/capecitabine
  * Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen
  * Known active or chronic hepatitis
* Medications

  * Currently or previously treated with angiopoietin inhibitors, or inhibitors of TIE-1 or TIE-2
  * Treatment with immune modulators such as cyclosporine or tacrolimus within 30 days prior to randomization
  * Treatment with sorivudine or its chemically related analogues
  * Anticoagulants (other than aspirin and anti-platelet agents) within 7 days prior to randomization. The concurrent use of low molecular weight heparin or heparanoids or low dose warfarin (i.e, ≤ 1 mg daily) for prophylaxis against thrombosis is acceptable while on study
* General

  * Not yet completed at least 30 days since ending other investigational device/drug trial(s), or subject is receiving other investigational treatments
  * Pregnant or is breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 22 months

SECONDARY OUTCOMES:
Safety and Tolerability | 22 months
Objective Response Rate (ORR) | 22 months
Duration of Response (DOR) | 22 months
Overall Survival (OS) | 22 months
Time to Progression (TTP) | 22 months
Time to Response | 22 months
Pharmacokinetics | 22 months
Patient Reported Outcomes | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Eatock MM, Tebbutt NC, Bampton CL, Strickland AH, Valladares-Ayerbes M, Swieboda-Sadlej A, Van Cutsem E, Nanayakkara N, Sun YN, Zhong ZD, Bass MB, Adewoye AH, Bodoky G. Phase II randomized, double-blind, placebo-controlled study of AMG 386 (trebananib) in combination with cisplatin and capecitabine in patients with metastatic gastro-oesophageal cancer. Ann Oncol. 2013 Mar;24(3):710-8. doi: 10.1093/annonc/mds502. Epub 2012 Oct 28. PMID 23108953
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com